CLINICAL TRIAL: NCT07096830
Title: Efficacy of Tetrachlorodecaoxide (TCDO) Drops in Chronic Wound Healing: Insights From a Randomized Controlled Trial
Brief Title: Efficacy of Tetrachlorodecaoxide (TCDO) Drops in Chronic Wound Healing
Acronym: TCDO-Wound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fazeelat Bibi (Other)
Responsible Party: Sponsor-Investigator, Fazeelat Bibi, General surgery resident, Khyber Teaching Hospital MTI-KTH Peshawar, Khyber Teaching Hospital
Organization: Khyber Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTH-RCT-TCDO-WOUND-2025-01
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Chronic Wound Care
MeSH Terms: interventions — tetrachlorodecaoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCDO + Standard Wound Care (Experimental): Participants in this group will receive topical Tetrachlorodecaoxide (TCDO, also known as Oxoferin®) drops applied directly to the wound bed once daily for 21 consecutive days, or until satisfactory healing is achieved. This will be administered alongside standard wound care practices, including saline irrigation, wound debridement, antibiotics as necessary, and sterile dressing.
  Interventions: Drug: Topical Tetrachlorodecaoxide (TCDO/Oxoferin); Other: Standard Wound Care
- Standard Wound Care Only (Active Comparator): Participants in this group will receive standard wound care practices, including saline irrigation, wound debridement, antibiotics as necessary, and sterile dressing, without the use of TCDO.
  Interventions: Other: Standard Wound Care

INTERVENTIONS:
Drug: Topical Tetrachlorodecaoxide (TCDO/Oxoferin) — Topical Tetrachlorodecaoxide (TCDO), a solution with antimicrobial and oxygen-releasing properties, will be applied once daily to the wound bed for 21 consecutive days or until satisfactory healing.
  Arms: TCDO + Standard Wound Care
Other: Standard Wound Care — Standard wound care includes saline irrigation, wound debridement, antibiotic administration as necessary, and sterile dressing. Provided to all participants.

SUMMARY:
This is a single-center, randomized controlled trial evaluating the effectiveness of topical tetrachlorodecaoxide (TCDO) solution in enhancing chronic wound healing. The study will compare standard wound care with and without the addition of topical TCDO drops. Eligible adult participants with chronic wounds of more than six weeks' duration will be randomly assigned to either the intervention or control group. The trial aims to assess the rate of wound healing, time to 50% wound closure, pain reduction measured by the Visual Analog Scale (VAS), and cost-effectiveness.

DETAILED DESCRIPTION:
Chronic wounds-including diabetic foot ulcers, arterial ulcers, venous leg ulcers, and pressure ulcers-represent a major clinical and economic burden in low-resource settings. Delayed healing increases the risk of infection, amputation, and prolonged hospitalization. Various topical agents have been used to enhance healing, with variable success. Tetrachlorodecaoxide (TCDO), a solution with antimicrobial and oxygen-releasing properties, has shown promising results in promoting granulation tissue. However, local clinical evidence is limited.

This randomized controlled trial aims to evaluate the effectiveness of topical tetrachlorodecaoxide (TCDO) in promoting chronic wound healing, compared to standard wound care alone. A total of 66 participants with chronic wounds (duration ≥ 6 weeks) will be enrolled in the Department of General Surgery, MTI Khyber Teaching Hospital (MTI-KTH), Peshawar. Participants will be randomly assigned to one of two groups: an intervention group receiving standard wound care plus topical TCDO application, or a control group receiving standard wound care alone. TCDO will be applied once daily (OD) for up to three weeks. Patients will be followed for up to 12 weeks to assess healing progress.

The primary outcome will be the percentage reduction in wound area, measured using the simple ruler method. Secondary outcomes include time to 50% wound closure, change in pain score using the Visual Analog Scale (VAS), wound Quality of Life (QoL) scores, and a cost-effectiveness analysis. Safety outcomes will be monitored throughout the study.

Ethical approval will be obtained from the MTI-KTH Institutional Review Board (IRB). The study will be conducted free of cost to participants and may offer an affordable treatment alternative to improve chronic wound care in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years diagnosed with chronic wounds (duration > 6 weeks)
* Wound size between 5 and 10 cm²
* Adequate perfusion:
* Ankle-Brachial Pressure Index (ABPI) > 0.8 for venous leg ulcers
* Palpable pulses for diabetic foot ulcers

Exclusion Criteria:

* Patients receiving immunosuppressive therapy or corticosteroids
* Presence of malignancy
* Patients who do not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in wound area (cm²) | Baseline to 4 weeks
  Wound area will be measured weekly using the simple ruler method by multiplying the longest length and the widest perpendicular width with a sterile ruler. The change in wound size from baseline to 4 weeks will be used to assess healing progress. A decrease in wound area will indicate improvement.

SECONDARY OUTCOMES:
Time to 50% wound closure | Baseline to 12 weeks
  Time (in days) required to achieve 50% reduction in wound area from the baseline measurement. Wound size will be assessed using the simple ruler method by multiplying the longest length and the widest perpendicular width. This outcome serves as an early indicator of treatment efficacy.
Change in pain score (Visual Analog Scale, VAS) | Baseline to 12 weeks
  Change in wound-related pain intensity assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain. Pain scores will be recorded at baseline and during follow-up visits to evaluate change in pain score over time.
Incidence of wound infection | Baseline to 12 weeks
  Incidence of clinical wound infection, determined by the presence of local signs of inflammation (e.g., redness, swelling, warmth), purulent discharge, or the need for antibiotic therapy as judged by the treating clinician.
Cost-Effectiveness of TCDO Treatment | Base line to 12 weeks
  Total treatment cost per patient will be compared between the intervention and control groups. Costs will include expenses related to wound dressings, hospital visits, medications, and other wound management components. This analysis will help determine the economic feasibility of using TCDO in resource-limited settings.
Change in wound-related quality of life (Wound-QoL) score | Base line to 12 weeks
  The impact of chronic wounds on patients' quality of life will be assessed using the validated Wound-Related Quality of Life (Wound-QoL) questionnaire. The Wound-QoL consists of 17 items, each scored from 0 to 4, resulting in a total score ranging from 0 (no impairment) to 68 (maximum impairment). Higher scores indicate worse quality of life. Scores will be measured at baseline and follow-up visits, and changes over time will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital, MTI KTH Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parikh R, Bakhshi G, Naik M, Gaikwad B, Jadhav K, Tayade M. The Efficacy and Safety of Tetrachlorodecaoxide in Comparison with Super-oxidised Solution in Wound Healing. Arch Plast Surg. 2016 Sep;43(5):395-401. doi: 10.5999/aps.2016.43.5.395. Epub 2016 Sep 21. PMID 27689045
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27689045/